CLINICAL TRIAL: NCT01856478
Title: A Randomised, Open-label, Phase III Study to Evaluate the Efficacy and Safety of Oral Afatinib (BIBW 2992) Versus Intravenous Methotrexate in Patients With Recurrent and/or Metastatic Head and Neck Squamous Cell Carcinoma Who Have Progressed After Platinum-based Therapy.
Brief Title: LUX-Head&Neck 3: Afatinib (BIBW2992) Versus Methotrexate for the Treatment of Recurrent and/or Metastatic Head and Neck Squamous Cell Cancer After Platinum Based Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1200.161; 1200-0161 (Other: Boehringer Ingelheim)
Record Dates: First submitted 2013-05-15; First posted 2013-05-17 (Estimated); Results first posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Head and Neck Neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Methotrexate; Afatinib

ARMS (2):
- Afatinib 40 mg (Experimental): Patients with recurrent and/or metastatic (R/M) head and neck squamous cell carcinoma (HNSCC) who progressed after being treated with platinum-based therapy took, orally, once daily one film-coated tablet of afatinib. Patients started with a 40 milligrams (mg) dose which could be escalated to 50 mg and/or reduced to 40 mg, 30 mg, or 20 mg, according to the absence of presence of drug-related adverse events (AEs).
  Interventions: Drug: Afatinib
- Methotrexate 40 mg (Active Comparator): Patients with recurrent and/or metastatic (R/M) head and neck squamous cell carcinoma (HNSCC) who progressed after being treated with platinum-based therapy received once weekly an intravenous bolus injection of methotrexate. Patients started with a 40 milligrams (mg) per square meter of body surface area (m^2) dose which could be escalated to 50 mg/m^2 and/or reduced to 40 mg/m^2, 30 mg/m^2, or 20 mg/m^2, according to the absence of presence of drug-related adverse events (AEs).
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Methotrexate — intravenous bolus injection once weekly
  Arms: Methotrexate 40 mg
Drug: Afatinib — oral intake of one film-coated tablet once daily
  Arms: Afatinib 40 mg

SUMMARY:
This randomized, open-label, phase III study will be performed in patients with recurrent and/or metastatic head and neck cancer which has progressed after platinum-based therapy. The objectives of this trial are to compare the efficacy and safety of afatinib versus methotrexate.

ELIGIBILITY:
Inclusion criteria:

* Histologically or cytologically confirmed squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx or larynx, which has recurred/metastasised and is not amenable for salvage surgery or radiotherapy.
* Documented progressive disease based on investigator assessment according to RECIST, following receipt of a cisplatin and/or carboplatin and/or Nedaplatin based regimen administered for recurrent and/or metastatic disease independent of whether patient progressed during or after platinum based therapy.
* Measurable disease according to RECIST (version 1.1).
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 at Visit 2.
* Male and female patients age is 18 years or older
* Signed and dated written informed consent that is in compliance with ICH-GCP and local law.

Exclusion criteria:

* Progressive disease within three months after completion of curatively intended treatment for locoregionally advanced or for metastatic head and neck squamous cell cancer (HNSCC).
* Primary tumour site nasopharynx (of any histology), sinuses, and/or salivary glands.
* Any other than one previous platinum based systemic regimen given for recurrent and/or metastatic disease, with the exception of immunotherapy used either before or after platinum based treatment. Re-challenge with the platinum based regimen after a temporary break is considered an additional line regimen only in case of progression within the break.
* Prior treatment with EGFR-targeted small molecules.
* Treatment with any investigational drug less than four weeks or anti-cancer therapy less than three weeks prior to randomization (except palliative radiotherapy to bones to alleviate pain).
* Unresolved chronic toxicity, other than hearing loss, tinnitus or dry mouth, CTCAE grade >2 from previous anti-cancer therapy or unresolved skin toxicities CTCAE grade >1 and/or diarrhoea CTCAE grade >1 caused by prior treatment with EGFR targeted antibodies.
* Previous tumour bleeding CTCAE grade =3.
* Requirement for treatment with any of the prohibited concomitant medications.
* Major surgical or planned procedure less than four weeks prior to randomization (isolated biopsies are not considered as major surgical procedures).
* Any other malignancy unless free of disease for at least five years except for:

  * Other HNSCC of a location as described in inclusion criterion number 1
  * Appropriately treated superficial basal cell skin cancer
  * Surgically cured cervical cancer in situ
  * For Korea: endoscopically cured superficial esophageal and/or gastric cancer is allowed
* Known lesion or signs of brain metastasis.
* Known pre-existing interstitial lung disease (ILD).
* Clinically relevant cardiovascular abnormalities, as judged by the investigator, such as, but not limited to, uncontrolled hypertension, congestive heart failure NYHA classification =III, unstable angina, myocardial infarction within six months prior to randomization, or poorly controlled arrhythmia.
* Significant or recent acute gastrointestinal disorders with diarrhoea as a major symptom in the opinion of the investigator, e.g. Crohn's disease, malabsorption or CTCAE grade >1 diarrhoea of any aetiology at randomization.
* Known HIV, active hepatitis B, active hepatitis C, and/or other known severe infections, including but not limited to tuberculosis, as judged by the investigator.
* Other significant disease that in the investigator's opinion would exclude the subject from the trial.
* Screening laboratory values:

  * Absolute neutrophil count (ANC) <1.5x10^9/l
  * Platelet count <75x10^9/l
  * Total bilirubin >1.5 times the upper limit of normal (ULN)
  * Aspartate amino transferase (AST) or alanine amino transferase (ALT) >3 times the ULN (if related to liver metastases >5 times the ULN)
  * Calculated creatinine clearance <50 ml/min (as evidenced by using the Cockcroft-Gault formula).
* Women of child-bearing potential and men who are able to father a child, unwilling to be abstinent or to use adequate contraception during the trial and for at least six months after end of treatment. Adequate methods of contraception and definition of child-bearing potential.
* Pregnancy or breast feeding.
* Known or suspected hypersensitivity to any of the study medications or their excipients.
* Patients unable to comply with the protocol, in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2013-06-07 (Actual); Primary Completion 2018-08-22 (Actual); Study Completion 2024-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (52):
- China (18):
  - Beijing Chao-Yang Hospital, Beijing
  - Cancer Hospital of Chinese Academy of Medical Science, Beijing
  - Navy General Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - The First Affiliated Hospital Of Bengbu Medical College, Bengbu
  - The First Hospital of Jilin University, Changchun
  - Sichuan Cancer Hospital, Chengdu
  - West China Hospital, Chengdu
  - Sun Yat-Sen University Cancer Center, Guangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - the 81th Hospital of PLA, Nanjing
  - Renji Hospital Shanghai Jiaotong Univesrity School of Medicine, Shanghai
  - Shanghai Changzheng Hospital, Shanghai
  - Shanghai Ninth People's Hospital, Shanghai
  - Fudan University Shanghai Cancer Center, Shanghai
  - Wuhan Union Hospital, Wuhan
  - Tongji Hospital, Tongji University, Wuhan
- Egypt (3):
  - Alexandria Clinical Research Center, Alexandria
  - National Cancer Institute, Cairo University, Cairo
  - Mansoura University Faculty of Medicine, Dakahlia
- Hong Kong (3):
  - Pamela Youde Nethersole Eastern Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
  - Prince of Wales Hospital, Shatin
- India (13):
  - Sujan Surgical Cancer Hospital, Amravati
  - Pristine Hospital, Bengaluru
  - Acharya Tulsi Regional Cancer Treatment & Research Institute, Bikaner
  - Rajiv Gandhi Government General Hospital, Chennai
  - M N J Institute of Oncology and Regional Cancer Centre, Hyderabad
  - Geetanjali Medical College and Hospital, Jaipur
  - J K Cancer Institute, Kanpur
  - B. P .Poddar Hospital & Medical Research Ltd., Kolkata, West Bengal
  - King George Medical University, Lucknow
  - Government Medical College & Hospital, Nagpur
  - Shatabdi Hospital, Nashik, Nashik
  - Ruby Hall Clinic, Pune
  - Noble Hospital Pvt Ltd, Pune
- Philippines (2):
  - Perpetual Succour Hospital (Cebu), Cebu City
  - St. Luke's Medical Center, Quezon City
- South Korea (5):
  - National Cancer Center, Goyang
  - Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St.Mary's Hospital, Seoul
  - Asan Medical Center, Seoul
- Taiwan (4):
  - Keelung Chang Gung Memorial Lover's Lake Branch, Keelung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Tri-Service General Hospital, Taipei
- Thailand (4):
  - Maharaj Nakom Chiangmai Hospital, Chiang Mai
  - Srinagarind Hospital, Muang
  - Naresuan University Hospital, Phitsanulok
  - Songklanagarind Hospital, Songkhla

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'.
  For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Guo Y, Ahn MJ, Chan A, Wang CH, Kang JH, Kim SB, Bello M, Arora RS, Zhang Q, He X, Li P, Dechaphunkul A, Kumar V, Kamble K, Li W, Kandil A, Cohen EEW, Geng Y, Zografos E, Tang PZ. Afatinib versus methotrexate as second-line treatment in Asian patients with recurrent or metastatic squamous cell carcinoma of the head and neck progressing on or after platinum-based therapy (LUX-Head & Neck 3): an open-label, randomised phase III trial. Ann Oncol. 2019 Nov 1;30(11):1831-1839. doi: 10.1093/annonc/mdz388. PMID 31501887
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Randomized, multicenter, open-label, active-control study with two parallel groups to investigate the efficacy and safety of afatinib versus methotrexate in patients with recurrent and/or metastatic (R/M) head and neck squamous cell carcinoma (HNSCC). Eligible patients were stratified by their Eastern Cooperative Oncology Group (ECOG) performance score and prior use of EGFR-targeted antibody therapy in the R/M. Patients were randomized to either afatinib or methotrexate in a 2:1 ratio.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Period: Overall Study
Arm/Group | Afatinib 40 mg | Methotrexate 40 mg
Started (Randomized) | 228 | 112
Treated | 228 | 104
Completed | 0 | 0
Not Completed | 228 | 112
Not completed — Not treated | 0 | 8
Not completed — Progressive disease per RECIST | 146 | 49
Not completed — Worsening of underlying cancer | 6 | 2
Not completed — Adverse events | 57 | 30
Not completed — Non-compliant with protocol | 1 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Refused to continue trial medication | 13 | 11
Not completed — Other reason than listed | 4 | 10

BASELINE CHARACTERISTICS:
Population: Randomized Set (RS): all patients who are randomized, regardless of taking investigational treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Afatinib 40 mg | Methotrexate 40 mg | Total
Number analyzed (Participants) | 228 | 112 | 340
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.7 (9.79) | 56.4 (9.36) | 55.2 (9.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 13 | 48
  Male | 193 | 99 | 292
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 215 | 107 | 322
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 13 | 5 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Secondary Outcome: Objective Response (OR)
Description: Objective response (OR) defined as the number of patients with best overall response of complete response (CR) or partial response (PR), according to RECIST 1.1. Complete response (CR) is defined as the disappearance of all target lesions and partial response (PR) is defined as decrease of at least 30% in the sum of the diameter of target lesions taking the baseline sum diameters as reference. Patients who did not show CR or PR were considered non-responders, irrespective of protocol violations or missing data.
Time Frame: From randomization until earliest of disease progression, death, or interim cut-off date (11-Apr-2019). Up to 35 months.
Population: Randomized Set (RS): all patients who are randomized, regardless of taking investigational treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Afatinib 40 mg | Methotrexate 40 mg
Number analyzed (Participants) | 228 | 112
Participants | 64 | 14
Statistical Analysis 1: Comparison: Afatinib 40 mg vs Methotrexate 40 mg; Stratified Cochran-Mantel-Haenszel was used to test the effect of afatinib compared with methotrexate. The stratification was done on the baseline ECOG performance score (0 or 1) and use of prior EGFR-targeted antibody in the R/M setting (Yes or No); Test type: Superiority; p = 0.0016, Cochran-Mantel-Haenszel — Null hypothesis: Afatinib and methotrexate have an equal response rate; Odds Ratio (OR) = 2.76, 95% CI 2-sided [1.47 to 5.18] — Linear regression stratified by baseline ECOG performance score and use of prior EGFR-targeted antibody in the R/M setting was used to calculate the OR of response and its confidence interval. Data presented as Afatinib versus Methotrexate

2. Primary Outcome: Progression Free Survival (PFS)
Description: Progression-free survival (PFS) was defined as the time from the date of randomization to the date of disease progression (PD) evaluated according to Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1 (v1.1). or to the date of death from any cause, whichever occurs first. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. PFS parameters were calculated based on Kaplan-Meier curves generated for each group.
Time Frame: From randomization until disease progression, death, or primary completion date, whichever occurs first. Up to 35 months.
Population: Randomized Set (RS): all patients who are randomized, regardless of taking investigational treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Afatinib 40 mg | Methotrexate 40 mg
Number analyzed (Participants) | 228 | 112
Months | 2.86 [2.79 to 3.71] | 2.56 [1.51 to 2.79]
Statistical Analysis 1: Comparison: Afatinib 40 mg vs Methotrexate 40 mg; Test type: Superiority — Stratified log-rank test was used to test the effect of afatinib on PFS compared with methotrexate. The stratification was done on the baseline ECOG performance score (0 or 1) and use of prior EGFR-targeted antibody in the R/M setting (Yes or No); p = 0.0005, Log Rank — Null hypothesis: Afatinib and methotrexate are equally effective in terms of PFS; Hazard Ratio (HR) = 0.627, 95% CI 2-sided [0.478 to 0.823] — Cox proportional hazards model stratified by baseline ECOG performance score and use of prior EGFR-targeted antibody in the R/M setting was used to calculate HR and its confidence interval. Data presented as Afatinib versus Methotrexate

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) defined as the time from the date of randomization to the date of death, regardless of its cause. OS parameters were calculated based on Kaplan-Meier curves generated for each group.
Time Frame: From randomization until death. Up to 6 years.
Population: Randomized Set (RS): all patients who are randomized, regardless of taking investigational treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Afatinib 40 mg | Methotrexate 40 mg
Number analyzed (Participants) | 228 | 112
Months | 6.93 [6.31 to 8.41] | 6.41 [5.16 to 8.38]
Statistical Analysis 1: Comparison: Afatinib 40 mg vs Methotrexate 40 mg; Stratified log-rank test was used to test the effect of afatinib compared with methotrexate. The stratification was done on the baseline ECOG performance score (0 or 1) and use of prior EGFR-targeted antibody in the R/M setting (Yes or No); Test type: Other; p = 0.3162, Log Rank; Hazard Ratio (HR) = 0.881, 95% CI 2-sided [0.687 to 1.129] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Time to Deterioration in Global Health Status
Description: Time to deterioration in global health status was defined as the time from randomization to the first decrease of 10 points on the global health/quality of life (QoL) scale. Patients with no deterioration (including those with disease progression) were censored at the last available health-related quality of life (HRQoL) assessment. The global health status (global health/QoL scale) was evaluated using the European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ-C30), a 30-item instrument designed to measure quality of life in cancer patients. It is composed of the overall health rating and the quality of life rating. The scale ranges from 0 to 100, where a higher score represents better global health status and quality of life.
Time Frame: From randomization until the earliest of deterioration, death, discontinuation with death within 4 weeks, or primary analysis date. Up to 30 months.
Population: Randomized Set (RS): all patients who are randomized, regardless of taking investigational treatment. Patients without global heath/quality of life scale values were excluded from the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Afatinib 40 mg | Methotrexate 40 mg
Number analyzed (Participants) | 217 | 104
Months | 4.17 [3.65 to 4.40] | 2.83 [2.63 to 7.75]
Statistical Analysis 1: Comparison: Afatinib 40 mg vs Methotrexate 40 mg; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.2121, Log Rank; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.54 to 1.15] — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Time to Deterioration in Pain Symptoms
Description: Time to deterioration in pain symptoms was defined as the time from randomization to the first decrease of 10 points on the pain scale. Patients with no deterioration (including those with disease progression) were censored at their last available health-related quality of life (HRQoL) assessment. The pain scale was evaluated using the pain module of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire for Head and Neck Cancer (EORTC QLQ-H&N35), which is designed to measure quality of life in head and neck cancer patients. It is composed of 4 questions, inquiring about pain in the mouth, pain in the jaw, soreness in the mouth, and a painful throat. The scale ranges from 0 to 100, where a higher score represents a higher symptom burden.
Time Frame: From randomization until the earliest of deterioration, death, discontinuation with death within 4 weeks, or primary analysis date. Up to 19 months.
Population: Randomized Set (RS): all patients who are randomized, regardless of taking investigational treatment. Patients without pain scale values were excluded from the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Afatinib 40 mg | Methotrexate 40 mg
Number analyzed (Participants) | 217 | 104
Months | 3.65 [3.02 to 4.40] | 2.96 [2.63 to 8.25]
Statistical Analysis 1: Comparison: Afatinib 40 mg vs Methotrexate 40 mg; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.9888, Log Rank; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.67 to 1.49] — [estimate comment as in outcome 2, analysis 1]

6. Secondary Outcome: Time to Deterioration in Swallowing
Description: Time to deterioration in swallowing was defined as the time from randomization to the first decrease of 10 points on the swallowing scale. Patients with no deterioration (including those with disease progression) were censored at their last available health-related quality of life (HRQoL) assessment. The swallowing scale was evaluated using the swallowing module of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire for Head and Neck Cancer (EORTC QLQ-H&N35), which is designed to measure swallowing difficulties in head and neck cancer patients. It is composed of 4 questions, inquiring about problems swallowing liquids, pureed food, solid food, and choking when swallowing. The scale ranges from 0 to 100, where a higher score represents greater difficulty in swallowing.
Time Frame: as for outcome 5
Population: Randomized Set (RS): all patients who are randomized, regardless of taking investigational treatment. Patients without swallowing scale values were excluded from the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Afatinib 40 mg | Methotrexate 40 mg
Number analyzed (Participants) | 216 | 104
Months | 4.11 [2.86 to 4.27] | 3.29 [2.56 to 7.39]
Statistical Analysis 1: Comparison: Afatinib 40 mg vs Methotrexate 40 mg; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.6260, Log Rank; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.62 to 1.34] — [estimate comment as in outcome 2, analysis 1]

7. Secondary Outcome: Change in Global Health Status Over Time
Description: Change in global health status over time was defined as the mean global health/QoL scale score up to the median follow-up time, describing the average global health status derived from the cumulative change over time, measured by the EORTC QLQ-C30. The EORTC QLQ-C30 is a 30-item questionnaire measuring quality of life in cancer patients (0 to 100, higher scores indicate better health/QoL).
  A mixed-effects growth curve model with a piecewise linear profile adjusted for baseline ECOG performance score and prior EGFR-targeted antibody use in R/M HNSCC was used. The change over time was calculated by dividing the area under the estimated growth curve (AUC) up to the median follow-up time by the median follow-up time.
  Timeframe: The model included measures at baseline and at the following timepoints, if available: Week 6, 12, 18, 24, 32, 40, 48, 56, 64, 72, 80, 88, 96, individual end of treatment (EOT; up to 36 months), and individual follow-up visit (EOT + 4 weeks, up to 37 months).
Time Frame: Mean change over time is reported up to 12 weeks. Detailed time frame in the endpoint description.
Population: Randomized Set (RS): all patients who are randomized, regardless of taking investigational treatment. Patients without post-baseline global heath/quality of life scale values were excluded from the analysis.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Afatinib 40 mg | Methotrexate 40 mg
Number analyzed (Participants) | 217 | 105
Units on a scale | 22.9 (3.53) | 15.0 (3.79)
Statistical Analysis 1: Comparison: Afatinib 40 mg vs Methotrexate 40 mg; Test type: Other; p = 0.0005, t-test, 2 sided; Adjusted mean difference = 7.9, 95% CI 2-sided [3.45 to 12.36] — Calculated as [Afatinib]-[Methotrexate]

8. Secondary Outcome: Change in Pain Scale Score Over Time
Description: Change in pain scale score over time was defined as the mean pain scale score up to the median follow-up time, describing the average pain score derived from the cumulative change over time, measured by the EORTC QLQ-H&N35 pain module. The EORTC QLQ-H&N35 pain module is a 4-question tool measuring pain in the mouth, jaw, throat, and soreness in the mouth (0 to 100, higher score = greater pain). A longitudinal mixed-effects growth curve model with a piecewise linear profile adjusted for baseline ECOG performance score and prior EGFR-targeted antibody use in R/M HNSCC was used. The change over time was calculated by dividing the area under the estimated growth curve (AUC) up to median follow-up time by the median follow-up time.
  Timeframe: The model included measures at baseline and at, if available: Week 6, 12, 18, 24, 32, 40, 48, 56, 64, 72, 80, 88, 96, individual end of treatment (EOT; up to 36 months), and individual follow-up visit (EOT + 4 weeks, up to 37 months).
Time Frame: Mean change over time is reported up to 12 weeks. Detailed time frame in the endpoint description.
Population: Randomized Set (RS): all patients who are randomized, regardless of taking investigational treatment. Patients without post-baseline pain scale values were excluded from the analysis.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Afatinib 40 mg | Methotrexate 40 mg
Number analyzed (Participants) | 217 | 105
Units on a scale | 7.6 (2.96) | 11.3 (3.39)
Statistical Analysis 1: Comparison: Afatinib 40 mg vs Methotrexate 40 mg; Test type: Other; p = 0.1090, t-test, 2 sided; Adjusted mean difference = -3.8, 95% CI 2-sided [-8.39 to 0.84] — Calculated as [Afatinib]-[Methotrexate]

9. Secondary Outcome: Change in Swallowing Scale Scores Over Time
Description: Change in swallowing scale score over time was defined as the mean swallowing scale score up to the median follow-up time, describing the average swallowing score derived from the cumulative change over time. It was assessed by EORTC QLQ-H&N35 swallowing module, a 4-question tool measuring problems swallowing liquids, pureed food, solid food, and choking when swallowing (0 to 100, higher score = greater difficulty swallowing). A longitudinal mixed-effects growth curve model with a piecewise linear profile adjusted for baseline ECOG and prior EGFR-targeted antibody use in R/M HNSCC was used. The change over time was calculated by dividing the area under the estimated growth curve (AUC) up to median follow-up time by the median follow-up time.
  Timeframe: the model included measures at baseline and at, if available: Week 6, 12, 18, 24, 32, 40, 48, 56, 64, 72, 80, 88, 96, individual end of treatment (EOT; up to 36 months), and individual follow-up visit (EOT + 4 weeks, up to 37 months)
Time Frame: Mean change over time is reported up to 12 weeks. Detailed time frame in the endpoint description.
Population: Randomized Set (RS): all patients who are randomized, regardless of taking investigational treatment. Patients without post-baseline swallowing scale values were excluded from the analysis.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Afatinib 40 mg | Methotrexate 40 mg
Number analyzed (Participants) | 216 | 105
Units on a scale | 10.1 (3.44) | 14.1 (3.85)
Statistical Analysis 1: Comparison: Afatinib 40 mg vs Methotrexate 40 mg; Test type: Other; p = 0.1819, t-test, 2 sided; Adjusted mean difference = -3.9, 95% CI 2-sided [-9.73 to 1.85] — Calculated as [Afatinib]-[Methotrexate]

10. Secondary Outcome: Number of Participants With Improvement in Pain Scale Score
Description: The number of participants with an improvement in pain scale scores is reported. Improvement was defined as a score that increases by at least 10 points (on a 0-100 point scale) from baseline at any time during the study. If a patient did not show improvement, worsening was defined as a 10-point decrease at any time during the study. Patients who neither improve nor worsen were considered stable. The pain scale was assessed using the pain module of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Head and Neck Cancer (EORTC QLQ-H&N 35). This questionnaire is designed to measure the quality of life in patients with head and neck cancer. It consists of four questions that inquire about pain in the mouth, pain in the jaw, soreness in the mouth, and a painful throat. The scale ranges from 0 to 100, where a higher score indicates a greater symptom burden.
Time Frame: Up to 37 months.
Population: Randomized Set (RS): all patients who are randomized, regardless of taking investigational treatment. Only patients with one baseline and one post-baseline results were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Afatinib 40 mg | Methotrexate 40 mg
Number analyzed (Participants) | 191 | 71
Participants
  Improved | 64 | 18
  Stable | 59 | 28
  Worsened | 68 | 25
Statistical Analysis 1: Comparison: Afatinib 40 mg vs Methotrexate 40 mg; Stratified logistic regression model stratified by baseline ECOG performance score (0 or 1) and use of prior EGFR-targeted antibody in the R/M setting (Yes or No) was used to compare the number of patients that of improved vs. not improved (i.e. stable and worsened) between the two treatment groups; Test type: Other; p = 0.222, Regression, Logistic; Odds Ratio (OR) = 1.46 — Afatinib versus Methotrexate

11. Secondary Outcome: Number of Participants With Improvement in Swallowing Scale Score
Description: The number of participants with an improvement in swallowing scale scores is reported. Improvement was defined as a score that increases by at least 10 points (on a 0-100 point scale) from baseline at any time during the study. If a patient did not show improvement, worsening was defined as a 10-point decrease at any time during the study. Patients who neither improve nor worsen were considered stable. The swallowing scale was assessed using the swallowing module of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Head and Neck Cancer (EORTC QLQ-H&N 35). This questionnaire is designed to measure swallowing difficulties in patients with head and neck cancer. It consists of four questions that inquire about problems swallowing liquids, pureed food, solid food, and choking when swallowing. The scale ranges from 0 to 100, where a higher score indicates greater difficulty in swallowing.
Time Frame: Up to 37 months.
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Afatinib 40 mg | Methotrexate 40 mg
Number analyzed (Participants) | 190 | 71
Participants
  Improved | 65 | 13
  Stable | 55 | 32
  Worsened | 70 | 26
Statistical Analysis 1: Comparison: Afatinib 40 mg vs Methotrexate 40 mg; [analysis description as in outcome 10, analysis 1]; Test type: Other; p = 0.012, Regression, Logistic; Odds Ratio (OR) = 2.37 — Afatinib versus Methotrexate

12. Secondary Outcome: Number of Participants With Improvement in Overall Health Rate of the Global Health Status
Description: The number of participants with an improvement in the overall health rate of global health status is reported. Improvement was defined as a score that increases by at least 10 points (on a 0-100 point scale) from baseline at any time during the study. If a patient did not show improvement, worsening was defined as a 10-point decrease at any time during the study. Patients who neither improve nor worsen were considered stable. The global health status (global health/QoL scale) was assessed using the European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ-C30), a 30-item instrument designed to measure quality of life in all cancer patients. It consists of the overall health rating and the quality of life rating. The scale ranges from 0 to 100, where a higher score indicates better global health status and quality of life.
Time Frame: Up to 37 months.
Population: Randomized Set (RS): all patients who are randomized, regardless of taking investigational treatment. Only patients with one baseline and one pos-baseline results were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Afatinib 40 mg | Methotrexate 40 mg
Number analyzed (Participants) | 191 | 71
Participants
  Improved | 92 | 21
  Stable | 33 | 19
  Worsened | 66 | 31
Statistical Analysis 1: Comparison: Afatinib 40 mg vs Methotrexate 40 mg; [analysis description as in outcome 10, analysis 1]; Test type: Other; p = 0.008, Regression, Logistic

13. Secondary Outcome: Number of Participants With Improvement in Quality of Life Rate of the Global Health Status
Description: The number of participants with an improvement in the quality of life rating of global health status is reported. Improvement was defined as a score that increases by at least 10 points (on a 0-100 point scale) from baseline at any time during the study. If a patient did not show improvement, worsening was defined as a 10-point decrease at any time during the study. Patients who neither improve nor worsen were considered stable. The global health status (global health/QoL scale) was assessed using the European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ-C30), a 30-item instrument designed to measure quality of life in all cancer patients. It consists of the overall health rating and the quality of life rating. The scale ranges from 0 to 100, where a higher score indicates better global health status and quality of life.
Time Frame: Up to 37 months.
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Afatinib 40 mg | Methotrexate 40 mg
Number analyzed (Participants) | 191 | 71
Participants
  Improved | 85 | 23
  Stable | 30 | 16
  Worsened | 76 | 32
Statistical Analysis 1: Comparison: Afatinib 40 mg vs Methotrexate 40 mg; [analysis description as in outcome 10, analysis 1]; Test type: Other; p = 0.091, Regression, Logistic

ADVERSE EVENTS:
Time Frame: All cause- mortality: From randomization until individual end of study. Up to 6 years. Adverse events reporting: From first drug administration until last drug administration, plus residual effect period. Up to approximately 6 years.
Description: All cause-mortality: Randomized Set (RS): all patients who are randomized, regardless of taking investigational treatment.
  Adverse event reporting: treated set: all randomised patients who were documented to have taken at least one dose of study medication.
Arm/Group | Afatinib 40 mg | Methotrexate 40 mg
All-Cause Mortality (participants affected / at risk) | 205/228 | 94/112
Serious Adverse Events (participants affected / at risk) | 90/228 | 36/104
Other Adverse Events (participants affected / at risk) | 217/228 | 89/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib 40 mg (N=228) | Methotrexate 40 mg (N=104)
Anaemia (Blood and lymphatic system disorders) | 5 | 3
Bone marrow failure (Blood and lymphatic system disorders) | 1 | 0
Bone marrow toxicity (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 2 | 0
Cardiac failure (Cardiac disorders) | 1 | 1
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 1 | 0
Eye swelling (Eye disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 9 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Gingival swelling (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 0
Asthenia (General disorders) | 3 | 2
Death (General disorders) | 4 | 2
Fatigue (General disorders) | 2 | 0
General physical health deterioration (General disorders) | 4 | 0
Localised oedema (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 4
Sudden cardiac death (General disorders) | 0 | 1
Sudden death (General disorders) | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 0 | 1
Liver injury (Hepatobiliary disorders) | 0 | 1
Abscess neck (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 3 | 0
Empyema (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Herpes virus infection (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 3 | 3
Oral infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 7 | 6
Respiratory tract infection (Infections and infestations) | 3 | 0
Sepsis (Infections and infestations) | 1 | 1
Septic shock (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 2 | 0
Soft tissue infection (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1
Tracheostomy malfunction (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 1
White blood cell count decreased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 4 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 0
Malnutrition (Metabolism and nutrition disorders) | 2 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 1 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Second primary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour compression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 2
Tumour inflammation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 2 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Coma (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Status epilepticus (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Completed suicide (Psychiatric disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 3
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1
Haemorrhage prophylaxis (Surgical and medical procedures) | 1 | 0
Circulatory collapse (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Shock (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib 40 mg (N=228) | Methotrexate 40 mg (N=104)
Anaemia (Blood and lymphatic system disorders) | 30 | 19
Leukopenia (Blood and lymphatic system disorders) | 1 | 16
Neutropenia (Blood and lymphatic system disorders) | 0 | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 6
Constipation (Gastrointestinal disorders) | 11 | 11
Diarrhoea (Gastrointestinal disorders) | 169 | 10
Mouth ulceration (Gastrointestinal disorders) | 28 | 6
Nausea (Gastrointestinal disorders) | 21 | 10
Stomatitis (Gastrointestinal disorders) | 44 | 11
Vomiting (Gastrointestinal disorders) | 26 | 5
Asthenia (General disorders) | 30 | 13
Fatigue (General disorders) | 20 | 15
Mucosal inflammation (General disorders) | 25 | 14
Pyrexia (General disorders) | 13 | 18
Paronychia (Infections and infestations) | 42 | 0
Alanine aminotransferase increased (Investigations) | 7 | 14
Aspartate aminotransferase increased (Investigations) | 6 | 11
Blood creatinine increased (Investigations) | 15 | 2
Haemoglobin decreased (Investigations) | 5 | 8
Neutrophil count decreased (Investigations) | 0 | 11
Platelet count decreased (Investigations) | 2 | 7
Weight decreased (Investigations) | 44 | 16
White blood cell count decreased (Investigations) | 7 | 12
Decreased appetite (Metabolism and nutrition disorders) | 32 | 12
Hypokalaemia (Metabolism and nutrition disorders) | 17 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 15 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 18 | 8
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 28 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 15 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 17 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 13 | 4
Rash (Skin and subcutaneous tissue disorders) | 100 | 8
Skin fissures (Skin and subcutaneous tissue disorders) | 12 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-01-03): https://cdn.clinicaltrials.gov/large-docs/78/NCT01856478/Prot_000.pdf
  • Statistical Analysis Plan (2016-04-01): https://cdn.clinicaltrials.gov/large-docs/78/NCT01856478/SAP_001.pdf